CLINICAL TRIAL: NCT01875627
Title: Comparing the Satiety Scores of a Carbohydrate Meal to a Meal of Equal Volume in Which Half of the Volume is Replaced With a Highly Viscous Gel.
Brief Title: Satiety Study of a Carbohydrate Meal to a Highly Viscous Gel Meal
Acronym: InGel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10-353
Record Dates: First submitted 2013-02-15; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Carbohydrate Noodles (Placebo Comparator): 0g Konjac Noodles
  Interventions: Dietary Supplement: Konjac noodles; Dietary Supplement: Carbohydrate and Konjac Noodles; Dietary Supplement: Carbohydrate noodles
- Carbohydrate and Konjac Noodles (Experimental): Half Carbohydrate and Half Non-Caloric Konjac Noodles - 122.5g Konjac
  Interventions: Dietary Supplement: Konjac noodles; Dietary Supplement: Carbohydrate and Konjac Noodles; Dietary Supplement: Carbohydrate noodles
- Konjac Noodles (Experimental): Non-Caloric Konjac Noodles (viscous gel meal) - 240g Konjac
  Interventions: Dietary Supplement: Konjac noodles; Dietary Supplement: Carbohydrate and Konjac Noodles; Dietary Supplement: Carbohydrate noodles

INTERVENTIONS:
Dietary Supplement: Konjac noodles — Replacement of carbohydrate noodles with non-caloric Konjac noodles (viscous gel meal)
  Other Names: Konnyaku - Konjac Noodles; Wellbond Import export; Scarborough, Ontario MIW 2P7
Dietary Supplement: Carbohydrate and Konjac Noodles
  Other Names: Konnyaku - Konjac Noodles; Wellbond Import export; Scarborough, Ontario MIW 2P7; Capellini n°1; Barilla America Inc.; Bannockburn, Il 60015
Dietary Supplement: Carbohydrate noodles
  Other Names: Capellini n°1; Barilla America Inc.; Bannockburn, Il 60015

SUMMARY:
To evaluate the effects of Konjac on satiety and subsequent food intake in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 18-65 years
* Having a BMI of 18.5 - 25 kg/m2
* No presence of major disease

Exclusion Criteria:

* Known history of liver or kidney disease, diabetes, hypertension, stroke or myocardial infarctions, thyroid disease, gastrointestinal disease, AIDS or AIDS-related complications; subjects using prescription medications or Natural Health Products; Subjects will be excluded if they have any condition which, in the opinion of the investigator, might jeopardize the health and safety of the subject or study personnel, or adversely affect the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Objective Satiety | 90 minutes
  Objective satiety will be measured through subsequent food intake.
  At each visit, participants will consume a pre-weighed snack (wafer cookies) that will be administered ad libitum at 90mins after consumption of the test meal. Subsequent food intake will be calculated by weighing the amount of the snack food left after consumption.

SECONDARY OUTCOMES:
Subjective Satiety | 90 minutes
  At each visit, participants will record their subjective satiety ratings using a 100 mm visual analogue scale and these rating will be combined into a total subjective appetite score using the formula (Q1+Q2+(100-Q3)+Q4)/4.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Risk Factor Modification Centre - St. Michael's Hospital
Locations (1):
- Risk Factor Modification Centre, Toronto, Ontario, Canada